CLINICAL TRIAL: NCT05065762
Title: Patient Preference for Treatment of Moderate-To-Severe Psoriasis in Japan
Brief Title: Measuring the Treatment Preferences of Participants in Japan With Moderate-to-Severe Psoriasis (PsO) Using Discrete Choice Experiment
Acronym: DCE
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-174
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Psoriasis
Keywords: Psoriasis; Japan; BMS-986165; Observational study; Moderate-to-severe PsO; DCE (discrete choice experiment); Preferences
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: Participants with moderate-to-severe Psoriasis (PsO) in Japan who have been recruited based on eligibility criteria
- Phase 2: Self-reported moderate-to-severe Psoriasis (PsO) participants in Japan

SUMMARY:
The purpose of this observational study is to identify and weight the treatment attributes from the moderate-to-severe Psoriasis (PsO) patients' perspective in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate-to-severe Psoriasis (PsO) by physician (phase 1) or self-reported (phase 2)
* Currently taking systemic psoriasis treatment
* Japanese resident aged 20 years and older

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Diagnosis of guttate, inverse, pustular, erythrodermic, or drug-induced psoriasis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 10 participants, diagnosed as moderate-to-severe Psoriasis (PsO) by a clinician were included in the Phase 1 qualitative interview
  A total of 200 participants, self-reported as moderate-to-severe PsO, were included in the Phase 2 online survey
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Psoriasis (PsO) patient preferences of moderate-to-severe systemic treatment atrribute | Within 60 minutes of survey/interview
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 1: Sex | At Baseline
Distribution of socio-demographic characteristics of PsO participants in Phase 1: Age | At Baseline
Distribution of clinical characteristics of PsO participants in Phase 1: Time since PsO diagnosis | At Baseline
Distribution of clinical characteristics of PsO participants in Phase 1: Severity of PsO | At Baseline
Distribution of clinical characteristics of PsO participants in Phase 1: Current treatments for PsO | At Baseline
Distribution of clinical characteristics of PsO participants in Phase 1: Time on current PsO treatment | At Baseline
Distribution of socio-demographic characteristics of PsO participants in Phase 1: Residence | At Baseline
Distribution of socio-demographic characteristics of PsO participants in Phase 1: Employment status | At Baseline
Distribution of socio-demographic characteristics of PsO participants in Phase 1: Education | At Baseline
Distribution of clinical characteristics of PsO participants in Phase 1: Total number of previous treatments | At Baseline
Distribution of clinical characteristics of PsO participants in Phase 1: Previous treatments for PsO | At Baseline
Distribution of socio-demographic characteristics of PsO participants in Phase 1: Level of income | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Sex | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Age | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Height | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Weight | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Residence | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Employment status | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Type of occupation | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Education | At Baseline
Distribution of clinical characteristics of Psoriasis (PsO) participants in Phase 2: Time since PsO diagnosis | At Baseline
Distribution of clinical characteristics of Psoriasis (PsO) participants in Phase 2: Self-reported severity | At Baseline
Distribution of clinical characteristics of Psoriasis (PsO) participants in Phase 2: Current treatments for PsO | At Baseline
Distribution of clinical characteristics of Psoriasis (PsO) participants in Phase 2: Time on current PsO treatment | At Baseline
Distribution of clinical characteristics of Psoriasis (PsO) participants in Phase 2: Previous treatments for PsO | At Baseline
Distribution of clinical characteristics of Psoriasis (PsO) participants in Phase 2: Comorbid conditions of interest | At Baseline
Distribution of socio-demographic characteristics of Psoriasis (PsO) participants in Phase 2: Level of income | At Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Morrisville, North Carolina, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm